CLINICAL TRIAL: NCT02853721
Title: Early Prediction of Hypocalcaemia Following Thyroid Surgery: A Prospective Randomized Clinical Trial
Brief Title: Early Prediction of Hypocalcaemia Following Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Alessandra Saba, Doctor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PG/2014/9514
Record Dates: First submitted 2016-05-06; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Hypocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): iPTH at 6 hours after surgery
  Interventions: Other: iPTH
- Control group (Other): no dosage of iPTH
  Interventions: Other: no dosage of iPTH

INTERVENTIONS:
Other: iPTH — iPTH assay six hours after surgery
  Arms: Experimental group
Other: no dosage of iPTH — Ca and P on postoperative day 1 and 2
  Arms: Control group

SUMMARY:
150 patients divided into two groups.The experimental group was submitted at the assay of iPTH six hours after surgery whilst the control group was submitted to a daily assay of serum calcium and phosphorus.

DETAILED DESCRIPTION:
Purpose: The aim of this randomized controlled trial was to validate the results of a previous prospective cohort study conducted in the same surgical unit regarding the use of concomitant intact parathyroid hormone (iPTH) and serum calcium measurement in predicting hypocalcemia after total thyroidectomy.

Methods: From January 2014 to January 2015, 150 patients underwent total thyroidectomy in our department and were divided into two groups. The experimental group was submitted at the assay of iPTH six hours after surgery whilst the control group was submitted to a daily assay of serum calcium and phosphorus. Sensitivity and specificity of different serum measurements have been calculated using the Receiver-operator characteristics (ROC) curve.

ELIGIBILITY:
Inclusion Criteria:

* Be submitted to total thyroidectomy during the study period
* Have signed the informed consent

Exclusion Criteria:

* Lack of inclusion criteria
* Lobectomy with isthmusectomy or partial or subtotal thyroidectomy
* Completion thyroidectomy
* Concomitant hyperparathyroidism was present
* Concomitant treatment with oral calcium and/or vitamin D prior to surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sensibility and specificity of iPTH and serum calcium measurement | 1 month
  Sensitivity and specificity of serum measurement using the Receiver-operator characteristics (ROC) curve

IPD SHARING:
Plan to Share IPD: Undecided